CLINICAL TRIAL: NCT01145365
Title: A Prospective Multicenter Trial Evaluating the Benefit of INitial Surgically Established Drainage Prior to Medical Therapy for the Treatment for Crohn's Perianal Fistulas
Brief Title: Study to Look at Benefit of Surgical Drainage Before Beginning Medical Therapy for Crohns Perianal Fistulas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Principal Investigator, David Schwartz, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100063
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Crohns Disease; Fistula; Abscess
Keywords: Crohns; Fistula; Perianal Abscess; Perianal
MeSH Terms: conditions — Crohn Disease; Fistula; Abscess

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination Therapy Group (Active Comparator): Patients in this arm will have surgically established drainage of their Crohns perianal fistulas and/or abscesses (exam under anesthesia (EUA)) done BEFORE beginning medical therapy with Cimzia.
  Interventions: Procedure: Exam under anesthesia (EUA)
- Control Group (No Intervention): Patients in this group will begin medical therapy with Cimzia regardless of status of surgically established drainage.

INTERVENTIONS:
Procedure: Exam under anesthesia (EUA) — EUA established drainage of perianal fistulas &/or abscesses will be done before patient begins medical therapy with certolizumab (Cimzia)
  Arms: Combination Therapy Group

SUMMARY:
This study is looking at the advantage of establishing surgical drainage for Crohn's fistulas and abscesses prior to starting medical therapy.

DETAILED DESCRIPTION:
Currently the importance of surgically established drainage of Crohn's perianal fistulas prior to medical therapy is controversial. Several retrospective studies have suggested a benefit to this approach. (1, 2) However, there have been no prospective studies performed to answer this important question. This study aims to definitively answer this question. Our hypothesis is that by establishing surgical drainage of all perianal fistulas and abscesses prior to initiation of medical therapy, further abscess formation will be prevented and the rate of durable fistula healing will improve.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female aged 18 years or older;
* A confirmed diagnosis of Crohn's disease and one or more identifiable perianal fistulas;
* Patient's standard of care treatment plan includes the following options: a) surgical intervention with an exam under anesthesia (EUA) by colorectal surgeon, seton placement and drainage of fistula prior to initiating Certolizumab or b) initiating Certolizumab without surgical intervention;
* Patient has had recent colonoscopy to determine disease activity and extent; and
* Patient has had either rectal EUS or pelvic MRI (type of test based on investigator site preference) which has identified one or more perianal fistulas.

Exclusion Criteria:

* Any of Inclusion Criteria is not met;
* Females who are pregnant or breast feeding;
* Anti-TNF use within 6 weeks prior to study entry;
* Patients who cannot take, or refuse to take concomitant immunosuppressive therapy with either azathioprine, 6-mercaptopurine, or methotrexate; Unless patient has been intolerant of these therapies in the past or is contraindicated as determined by the investigator.
* Patients who cannot take, or refuse to take concomitant antibiotic therapy;
* Patients with severe anal stenosis or tenderness which would preclude colonoscopy and / or rectal EUS;
* Patients who cannot take or refuse to take certolizumab;
* Patients with active or latent tuberculosis;
* Patients who have had systemic antibiotic, antiviral or antifungal treatment(s) within 3 weeks prior to Screening for all non-Crohn's related infections;
* Patients concurrently taking anakinra (Kineret);
* Patients with a history of cancer or lymphoproliferative disease other than a successfully and completely treated cutaneous squamous cell or basal cell carcinoma or carcinomain-situ of the cervix;
* Patients with chronic hematologic problems such as bleeding dyscrasias;
* Patients with a history of demyelinating disease (i.e. multiple sclerosis); and
* Patients with congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Surgical drainage of all perianal fistulas & abscesses prior to start of medical tx improves rate of healing & prevents further abscess formation. | 54 weeks
  Our hypothesis is that by establishing surgical drainage of all perianal fistulas and abscesses prior to initiation of medical therapy, further abscess formation will be prevented and the rate of durable fistula healing will improve.

CONTACTS AND LOCATIONS:
Overall Officials: David A Schwartz, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (3):
- United States (3):
  - University of Maryland, Baltimore, Maryland
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee